CLINICAL TRIAL: NCT03888144
Title: Study of Ketorolac Versus Opioid for Pain After Endoscopy (SKOPE): A Double-blinded Randomized Control Trial Comparing Outpatient Analgesic Efficacy of NSAIDs and Opioids in Patients Undergoing Ureteroscopy for Kidney Stones
Brief Title: Study of Ketorolac Versus Opioid for Pain After Endoscopy
Acronym: SKOPE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-872
Record Dates: First submitted 2019-03-14; First posted 2019-03-25 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Kidney Calculi; Ureteral Calculi
MeSH Terms: conditions — Kidney Calculi; Ureteral Calculi | interventions — Oxycodone; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxycodone group (Active Comparator): Patients randomized to 20 pills of 5 mg oxycodone by mouth every 6 hours as needed for pain after ureteroscopy.
  Interventions: Drug: Oxycodone
- Ketorolac group (Experimental): Patients randomized to 20 pills of 10 mg ketorolac by mouth every 6 hours as needed for pain after ureteroscopy.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Oxycodone — 5 mg of oxycodone taken by mouth every 6 hours for 5 days
  Arms: Oxycodone group
Drug: Ketorolac — 10 mg of ketorolac taken by mouth every 6 hours for 5 days
  Other Names: Toradol
  Arms: Ketorolac group

SUMMARY:
A double blind randomized controlled trial designed to compare pain control and safety with ketorolac and oxycodone in the post-operative setting for patients undergoing ureteroscopy for treatment of urinary stones. Patients are followed for five days after their surgery as they record their pain scores, medication utilization, and stent related symptoms.

DETAILED DESCRIPTION:
Pain is the leading cause for unplanned emergency department visits and readmissions after ureteroscopy (URS), making post-operative analgesic stewardship a priority given the current opioid epidemic. The investigators conducted a double-blinded, randomized controlled trial (RCT), with non-inferiority design, comparing nonsteroidal anti-inflammatory drugs (NSAIDs) to opiates for postoperative pain control in patients undergoing URS for urolithiasis.

Patients were randomized and blinded to either oxycodone (5mg) or ketorolac (10mg), taken as needed, with 3 non-blinded oxycodone rescue pills for breakthrough pain. Primary study outcome was visual analog scale pain score on post-operative days 1-5. Secondary outcomes included medication utilization, side effects, and Ureteral Stent Symptoms Questionnaire (USSQ) scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients with kidney or ureteral stones confirmed on imaging (CT of the abdomen pelvis) and who elect for definitive treatment via unilateral ureteroscopy at one of two hospital sites within a tertiary care institution
* Patients who post-operatively receive a unilateral ureteral stent
* Capable of giving informed consent
* Capable and willing to fulfill requirements of the study

Exclusion Criteria:

* Active or history of peptic ulcer disease, gastrointestinal bleeding or perforation
* History of coronary artery bypass graft surgery
* History of a bleeding disorder
* GFR less than 60 mL/min/1.73m2 (MDRD equation)
* Chronic use of opioid or other pain medication including NSAIDs (greater than 12 weeks)
* Known allergy to either ketorolac or oxycodone
* Known or suspected pregnancy
* Solitary kidney
* Patients taking anticoagulant medication or antiplatelet medication (e.g. warfarin, clopidogrel, pradaxa, rivaroxaban, apixaban etc).
* Inability to give informed consent or unable to meet requirements of the study for any reason

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sriharan Sivalingam, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxycodone Group | Ketorolac Group
Started | 43 | 38
Completed | 43 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxycodone Group | Ketorolac Group | Total
Number analyzed (Participants) | 43 | 38 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 38 | 81
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (14.0) | 53.8 (12.4) | 52.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 16 | 40
  Male | 19 | 22 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 38 | 33 | 71
  Non Caucasian | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Pain Score
Description: Patient Reported Visual Analogue Score scored from 0-10 with lower scores equaling less pain.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxycodone Group | Ketorolac Group
Number analyzed (Participants) | 43 | 38
units on a scale | 4.6 (3.1) | 4.5 (2.9)

2. Secondary Outcome: Number of Study Pills Used
Description: the use of opioid medication as per the study protocol; Required study pills
Time Frame: Post-operative days 1 to 5
Population: 5 patients in the Oxy group and 2 in the Ketorolac group didn't require meds so they were excluded from final calculation
Measure: Mean (Standard Deviation); unit: number of pills used
Arm/Group | Oxycodone Group | Ketorolac Group
Number analyzed (Participants) | 38 | 36
number of pills used | 7.3 (6.1) | 7.1 (5.2)

3. Secondary Outcome: Use of Rescue Medication (Opioid)
Description: the use of rescue opioid medication as per the study protocol; use of rescue medication by the patients
Time Frame: post operative day 1-5
Population: not all enrolled subjects used rescue medications
Measure: Mean (Standard Deviation); unit: number of pills used
Groups:
- Oxycodone Group; Ketorolac Group: Patients were randomized and blinded to either oxycodone (5 mg) or ketorolac (10 mg), taken as needed, with 3 nonblinded oxycodone rescue pills for breakthrough pain
Arm/Group | Oxycodone Group | Ketorolac Group
Number analyzed (Participants) | 21 | 11
number of pills used | 1.1 (1.3) | 0.8 (1.2)

4. Other Pre Specified Outcome: Day in Bed
Description: number of days patient spent confined to bed post operatively
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Oxycodone Group | Ketorolac Group
Number analyzed (Participants) | 41 | 38
days | 2.3 (2.6) | 1 (1.3)

5. Other Pre Specified Outcome: Visual Analogue Scale (VAS)
Description: VAS as reported by the patients while in PACU (score from 0-10, with 0 meaning no pain and 10 max pain)
Time Frame: Up to 5 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oxycodone Group | Ketorolac Group
Number analyzed (Participants) | 41 | 38
units on a scale | 4.6 (3.1) | 4.5 (2.9)

ADVERSE EVENTS:
Time Frame: the side effects have been reported over the study period of 2 years
Arm/Group | Oxycodone Group | Ketorolac Group
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/38
Other Adverse Events (participants affected / at risk) | 12/43 | 11/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone Group (N=43) | Ketorolac Group (N=38)
nausea (Gastrointestinal disorders) | 12 (12) | 11 (11) — patient felt nausea and impending vomiting
vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) — patient who had actual vomiting as a medication side effect

LIMITATIONS AND CAVEATS:
This study has limitations: medication adherence and symptom scores relied on self-reporting; some patients had early stent removal or were lost to follow-up; the population excluded sicker patients; and most were Caucasian at a tertiary center, limiting generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT03888144/Prot_SAP_000.pdf